CLINICAL TRIAL: NCT01456715
Title: Immunogenicity and Safety of Gardasil and Twinrix Vaccines Co-administered or Administered a Month Apart, According to the 0, 6 Months Schedule and the Effect of a Third Dose of Gardasil or Cervarix Administered 42 Months Later.
Brief Title: Immunogenicity of Gardasil and Twinrix and the Effect of a Dose of Gardasil or Cervarix Given 42 Months Later.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Vladimir Gilca, Principal investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 122.05.01; 9427-L1802/1-21C (Other: Health Canada)
Record Dates: First submitted 2011-10-18; First posted 2011-10-21 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Human Papillomavirus
Keywords: Human Papillomavirus Vaccines; Immunogenicity Gardasil Cervarix; Booster dose
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gardasil, Immunogenicity, Booster dose. (Active Comparator)
  Interventions: Biological: Gardasil vaccine, Immunogenicity, Booster dose.
- Cervarix, Immunogenicity, Booster dose. (Experimental)
  Interventions: Biological: Cervarix Vaccine, Immunogenicity, Booster Dose.

INTERVENTIONS:
Biological: Gardasil vaccine, Immunogenicity, Booster dose. — Gardasil vaccine given according to the 0,6 months schedule and a booster dose of Gardasil given 42 months later.
  Other Names: HPV vaccine
  Arms: Gardasil, Immunogenicity, Booster dose.
Biological: Cervarix Vaccine, Immunogenicity, Booster Dose. — Gardasil vaccine given according to the 0,6 months schedule and a booster dose of Cervarix given 42 months later.
  Other Names: HPV vaccine.
  Arms: Cervarix, Immunogenicity, Booster dose.

SUMMARY:
Two human papillomavirus vaccines are now commercially available.

No clinical data exist regarding:

* The immunogenicity and safety of Gardasil and Twinrix when co-administered.
* The immunogenicity and safety of Cervarix when administered to subjects previously vaccinated with Gardasil.

The main objective of the first phase of this clinical trial was:

• To assess and compare the immunogenicity of Gardasil and Twinrix Junior when co-administered or administered at one month interval according to a 0, 6 month schedule to 9-10 year-old girls.

The main objective of the seconde phase of this clinical trial is:

• To determine the effect of a booster dose of Gardasil or Cervarix on HPV antibodies when given 42 months post-vaccination of 9-10 year-old girls with two doses of Gardasil.

Study Design & Duration:

Experimental Design: Blind for the third HPV vaccine dose, randomized, single centre study with two treatment groups.

Duration of the study:

Participants will be followed for the duration of 10 years post-primary vaccination.

Number of Centres:

One Center.

ELIGIBILITY:
Inclusion Criteria:

* In 2008-2009 received two doses of Gardasil at the age of 9-10 years according to 0, 6 months schedule.

Exclusion Criteria:

* Received less than two doses of Gardasil or received an HPV vaccine outside the study protocol.

Ages: 12 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 418 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Antibody to HPV | 1 month post booster dose
  The effect of a booster dose of Gardasil or Cervarix administered randomly (1:1) to subjects vaccinated 42 months before with two doses of Gardasil.

SECONDARY OUTCOMES:
Safety of a booster dose of Gardasil and Cervarix administered 42 months after the second dose of Gardasil. | Solicited adverse events 5 days post vaccine administration. Serious adverse events during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Gilca, MD, PhD, Principal Investigator — INSPQ, CHUQ-CHUL, Laval University
Locations (1):
- Laval University Research Hospital Center, Québec, Canada